CLINICAL TRIAL: NCT01188200
Title: Four-Hour Evaluation of a Medical Food in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Bobbie Swearengin, Director Clinical Research, Abbott Nutrition
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BK79
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2010-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutritional Formula #M979 (Experimental): nutritional formula
  Interventions: Other: Experimental nutritional formula #M979
- Regular standard meal (Active Comparator): standard meal
  Interventions: Other: Standard food

INTERVENTIONS:
Other: Experimental nutritional formula #M979 — One two hundred and forty mL serving at test time, taken orally
  Arms: Nutritional Formula #M979
Other: Standard food — Standard meal prior to test time
  Arms: Regular standard meal

SUMMARY:
The purpose of this study is to demonstrate the efficacy of a nutritional formula in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has type 2 diabetes.
2. Subject is over 18 years of age.
3. Subject is a male, or a non-pregnant, non-lactating female.
4. Subject's BMI is > 20 kg/m2 and < 40 kg/m2.
5. Subject's HbA1c level is 6.5 - 11%.
6. If on a chronic thyroid medication or hormone replacement therapy, subject has been on constant dosage for at least two months prior to Screening Visit.
7. Subject's weight is stable for the past two months prior to Screening Visit.

Exclusion Criteria:

1. Subject uses exogenous insulin, Byetta or alpha-glucosidase inhibitor for glucose control.
2. Subject has type 1 diabetes.
3. Subject has history of diabetic ketoacidosis.
4. Subject has the following: current infection ; has had inpatient surgery or received systemic corticosteroid treatment in the last 3 months; or antibiotics in the last 3 weeks prior to screening.
5. Subject has an active malignancy.
6. Subject has had significant cardiovascular event <6 months prior to study entry or history of congestive heart failure.
7. Subject has end stage organ failure.
8. Subject has history of severe gastroparesis, renal or hepatic disease.
9. Subject has an active metabolic, hepatic, or gastrointestinal disease or condition that may interfere with nutrient absorption, distribution, metabolism, or excretion, excluding diabetes.
10. Subject has a chronic, contagious, infectious disease.
11. Taking daily medications at doses that would interfere with nutrient absorption, metabolism, excretion, gastric motility, or blood glucose.
12. Subject has fainted or experienced other adverse event in response to blood collection prior to enrollment into this study.
13. Clotting or bleeding disorders.
14. Allergic or intolerant to any ingredient found in the test meal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2009-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The primary variable is glucose concentration | 0 to 240 minutes

SECONDARY OUTCOMES:
Additional measures of glucose concentration | 0 to 240 mins

CONTACTS AND LOCATIONS:
Overall Officials: Anne Voss, PhD, Study Chair — Abbott Nutrition
Locations (11):
- Russia (11):
  - Kuban State Medical University, Krasnodar
  - City Clinical Hospital #68, Moscow
  - City Clinical Hospital #52, Moscow
  - City Hospital #67, Moscow
  - Novosibirsk State Medical University, Novosibirsk
  - State Novosibirsk Regional Hospital, Novosibirsk
  - City Clinical Hospital #3, Saint Petersburg
  - Medical Centre Twenty First Century, Saint Petersburgh
  - Diabetes Centre, LLC, Samara
  - Tyumen State Medical Academy, Tyumen
  - Bashkir State Medical University, Ufa